CLINICAL TRIAL: NCT05664412
Title: Using Transcranial Alternating Current Stimulation With Starstim Home Device to Improve Executive Function in Youths With 22q11.2 Deletion Syndrome: A Randomized Double-blind Sham-controlled Study
Brief Title: Using Transcranial Alternating Current Stimulation to Improve Executive Function in 22q11.2 Deletion Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stephan Eliez (Other)
Responsible Party: Sponsor-Investigator, Stephan Eliez, Professor, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-D0123
Record Dates: First submitted 2022-12-06; First posted 2022-12-23 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: 22Q11 Deletion Syndrome; tACS
MeSH Terms: conditions — 22q11 Deletion Syndrome

STUDY DESIGN:
Intervention Model Description: This is a randomized double-blind sham-controlled study. We will use transcranial alternating current stimulation (tACS) of the dorsolateral prefrontal cortex and temporal cortex by adopting a high-density (HD) montage with 3 electrodes to target the dorsolateral prefrontal cortex and 3 electrodes to target the temporal cortex. To select individualized parameters for stimulation, we will first acquire and analyse structural MRI (comprising T1 and T2-weighted sequences) and EEG data during a working memory task. The first arm will receive one session of HD-tACS per day for 5 consecutive days every week over four weeks; each session will last 21 minutes. All sessions will occur during cognitive training (i.e., execution of a working memory task). The second arm will first receive 20 sessions of sham stimulation coupled with cognitive training. After the one-month follow-up, they will receive in-phase offline theta tACS (i.e., tACS at rest, with no task).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Care providers, outcome assessors, data analysts, and a research assistant who will follow the procedures remotely will be blind. A person in the lab not directly involved in any of the previously mentioned activities will be aware of the randomization for safety reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): Participants will receive 20 sessions of In-phase online theta tACS paired with working memory training.
  Interventions: Device: at-home tACS using Starstim-Home tES
- Control group (Sham Comparator): Participants will receive 20 sessions of sham tACS paired with working memory training. After unblinding (by someone from our lab but external to the study), they will receive 20 sessions of in-phase offline theta tACS.
  Interventions: Device: at-home tACS using Starstim-Home tES

INTERVENTIONS:
Device: at-home tACS using Starstim-Home tES — We will use transcranial alternating current stimulation (tACS) of the dorsolateral prefrontal cortex and temporal cortex by adopting a high-density (HD) montage with 3 electrodes to target the dorsolateral prefrontal cortex and 3 electrodes to target the temporal cortex. To select individualized parameters for stimulation, we will first acquire and analyse structural MRI (comprising T1 and T2-weighted sequences) and EEG data during a working memory task. We planned one session of HD-tACS per day for 5 consecutive days every week over four weeks; each session will last 21 minutes. All sessions will occur during cognitive training (i.e., execution of a working memory task).

SUMMARY:
The purpose of this project is to explore the effects of transcranial alternating current stimulation (tACS) in children, adolescents and young adults with a 22q11.2 microdeletion. The main aim of the present research project is to investigate the effects of repeated, individually tuned high-density (HD) tACS on cognition (i.e., WM performance) and related neuroimaging markers in carriers of the 22q11DS. As cognitive deficits, most notably WM impairment, are among the earliest signs of psychotic disorders, interventions during adolescence aimed at reducing cognitive decline in at-risk individuals may prove effective in delaying or even preventing the later emergence of psychotic symptoms.

DETAILED DESCRIPTION:
22q11.2 is the neurogenetic disorder with the highest genetic risk of schizophrenia and early diagnosis allows subjects to be followed from early childhood. Not only does atypical cognitive development precede the emergence of the first psychotic symptoms, but it predicts their later severity and further cognitive decline. Even in subjects which premorbid cognitive functioning is already low due to neurogenetic syndromes, further decline in cognitive abilities indicates an increased risk for the emergence of psychotic symptoms.

psychotic symptoms. Thus, early intervention targeting cognition could potentially mitigate the burden of the disease. Individuals carrying the 22q11.2 microdeletion have a distinctive cognitive profile characterized by a dissociation between verbal and visual-spatial memory capacities, supporting a specific deficit in the processing of visuo-spatial information. Memory deficits are therefore a specific weakness of this population. For this reason, we designed a non-invasive brain stimulation protocol to improve visual working memory (WM) in adolescents and young adults with 22q11DS using individual parameters to account for age individual parameters to account for participant age and anatomical variability.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed genetic diagnosis of 22q11DS
* Age between 14 and 25 years old
* Willingness to participate
* Informed Consent signed by the subject and/or the caregiver(s)

Exclusion Criteria:

* Epilepsy
* Deep brain stimulation electrodes
* Traumatic brain injury
* Facial metal implants

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of adverse events following tACS (safety and tolerability) | 1 month (i.e., duration of 20 tACS sessions)
  Safety and tolerability of using at-home stimulation in a group of youths with neurodevelopmental disorders (i.e., 22q11DS) with the help of caregivers. It will be measured using a homemade questionnaire assessing the presence and intensity of side effects of tACS (e.g., headache, tingling, skin redness, neck pain). Each side effect will be rated on a intensity scale from 1 (absent) to 4 (severe). In addition, we will assess whether the side effect is associated with tACS, from 1 (no association) to 5 (certain association). This questionnaire is present in the Clinical Report Form (CRF) and will be filled after each stimulation session (both tACS and sham stimulation).

SECONDARY OUTCOMES:
Change in verbal working memory performance using Digit Span subtest (Weschler's child/adult intelligence scale (2004, 2011). | An average of 3 months (i.e., duration of the study protocol)
  We will investigate whether there is a direct positive effect of tACS on verbal working memory using parallel versions of Digit Span (forward, reverse, and sequencing conditions) inspired Weschler's child/adult intelligence scale (Weschler, 2004, 2011). This will be assessed at three visits: baseline (i.e., pre-stimulation), post-stimulation, 1-month follow-up.
Change in visuospatial working memory performance using Leiter-3 scales (Roid, Mille, Pomplun, & Koch, 2013), Testing of Attentional Performance (Zimmermann & Fimm, 2002), and CANTAB software (Cambridge Cognition, 2019) | An average of 3 months (i.e., duration of the study protocol)
  We will investigate whether there is a direct positive effect of tACS on visual working memory using parallel versions of Forward memory and Reverse memory subtests, inspired from Leiter-3 (Roid, Mille, Pomplun, & Koch, 2013) and visual n-back task from Testing of Attentional Performance (Zimmermann & Fimm, 2002), and Spatial Working Memory from CANTAB (Cambridge Cognition, 2019). This will be assessed at three visits: baseline (i.e., pre-stimulation), post-stimulation, 1-month follow-up.
Change in the oscillatory response of the brain related to working memory with EEG using time-frequency + cross-frequency coupling analyses | An average of 3 months (i.e., duration of the study protocol)
  Using a visual working memory EEG task, we will explore the oscillatory response of the brain related to working memory. For the EEG analyses, we will use a pipeline that has already been applied to previous data and described in detail (Mancini, Rochas, Seeber, Grent-'t-Jong, et al., 2022a; Mancini, Rochas, Seeber, Roehri, et al., 2022b). All participants will do one EEG at each visit (baseline, post-stimulation, 1-month follow-up).
Change in psychotic experiences using Ecological Momentary Assessment (EMA) | An average of 3 months (i.e., duration of the study protocol)
  Participants will complete a EMA protocol for approximately 3 months (one notification per day). The protocol will be implemented on the RealLife Exp app, developed for clinical research purposes. The data is encrypted at rest and its transmission is secured using several different methods. The data will be transferred on the server of the University of Geneva. Participants will complete the EMA questionnaire once they hear a notification. A follow-up call will be scheduled with the participant to ensure compliance. At each beep, psychotic experiences will be assessed using a series of items (e.g. " Seeing or hearing things others don't perceive ") rated on a 7-point Likert scale (1 = " not at all " to 7 = " extremely "). Feller et al. (2021) showed an association between psychotic experiences (measured by EMA) and severity of psychotic symptoms (measured by a gold standard assessment) in 22q11DS. Their study shows feasibility and validity of assessing psychotic experiences with EMA.
Change in Attention-Deficit/Hyperactivity Disorder (ADHD) symptoms using EMA | An average of 3 months (i.e., duration of the study protocol)
  Details about storage and security of EMA data can be found in Secondary Outcome 5. The EMA questionnaire will include other items, regarding ADHD symptoms. At each beep, ADHD symptoms will be assessed using a series of items (e.g. " Being easily distracted ") rated on a 7-point Likert scale (1 = " not at all " to 7 = " extremely ").

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Latreche C, Mancini V, McGinn N, Rochas V, Ferat V, Forrer S, Schneider M, Eliez S. Safety and feasibility of home-based transcranial alternating current stimulation in youths with 22q11.2 deletion syndrome. Front Neurosci. 2024 Oct 24;18:1453839. doi: 10.3389/fnins.2024.1453839. eCollection 2024. PMID 39513044